CLINICAL TRIAL: NCT04355780
Title: Immunologic Features of Respiratory Failure in Pediatric Hematopoietic Cell Transplantation (HCT) Recipients and Pediatric Oncology Patients
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HCTALI
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Failure; Respiratory Disease
MeSH Terms: conditions — Respiratory Insufficiency; Respiration Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subgroup 1: Composed of HCT patients with respiratory failure requiring intubation and mechanical ventilation.
- Subgroup 2: Composed of oncology patients (solid tumor or leukemia patients) who have not undergone HCT and who have respiratory failure requiring intubation and mechanical ventilation.
- Subgroup 3: Composed of chimeric antigen T-cell receptor infusion recipients who have respiratory failure requiring intubation and mechanical ventilation.

SUMMARY:
This study is being done because researchers want to learn more about genes that control the immune response in the participant's lungs and blood when the participant have lung disease leading to respiratory failure.

Primary Objective

To evaluate the feasibility of performing single cell gene expression analyses on tracheal aspirates from immunocompromised pediatric patients with immune compromising conditions, including HCT recipients.

Secondary Objectives

* To assess whether cell composition and activation states in longitudinally obtained tracheal aspirate and blood samples are able to distinguish unique immunopathology for each of the early post-HCT lung diseases.
* To assess whether cell composition and activation states in longitudinally obtained tracheal aspirate and blood samples are different between two immunodeficient patient populations (alloHCT vs non alloHCT) with lung disease and respiratory failure.
* To test the hypothesis that allogeneic T cell responses are implicated in the pathogenesis of early post-HCT lung diseases.

Exploratory Objectives

To correlate immune cell signaling in the lower respiratory tract and blood of patients with early post-HCT lung diseases with the presence or absence of pathogenic microbes at each site.

To explore HLA testing in Tracheal Aspirates in samples where enough cells are present.

DETAILED DESCRIPTION:
This study involves a Tracheal aspirate, Bronchoalveolar lavage (BAL), and blood samples. The tracheal aspirates and blood samples will be obtained within 24 hours of intubation, then twice more every 3 -4 days, and then once a week until the patient is extubated. If the primary treatment team performs bronchoscopy with BAL, then an aliquot of residual BAL fluid will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Participant is age 0 to 21 years old
* Participant has acute respiratory failure due to primary pulmonary disease and is expected to receive invasive mechanical ventilation for more than 48 hours

Exclusion Criteria:

* The primary etiology of respiratory failure is not related to primary pulmonary disease
* Aspiration is present
* The participant has a tracheostomy
* If the patient has undergone HCT, they are more than 100 days removed from HCT
* Has a diagnosis of severe combined immunodeficiency syndrome (SCIDS)
* The primary on-service team feels obtaining a study sample would be unsafe for any reason.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All participants who meet eligibility criteria and consent to enrollment on the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of performing single cell gene expression analyses on tracheal aspirates | 4 years
  Feasibility is a qualitative binary outcome (Yes and No), based on the success of recovery of more than 100,000 live cells from a tracheal aspirate and blood sample from five of the first ten allo HCT patients enrolled on the study protocol.

SECONDARY OUTCOMES:
Success of distinguishing unique immunopathology for each of the early post-HCT lung diseases | 4 years
  This is a qualitative binary outcome (Yes/No) by applying single cell gene expression analyses to cells from tracheal aspirates and blood of patients with post-HCT lung diseases. With visualization techniques, a call of success (Yes/No) will be made.
: Difference of cell composition and activation states between two immunodeficient patient populations (alloHCT vs non alloHCT) with lung disease and respiratory failure. | 4 years
  This is a qualitative binary outcome (different vs not different) obtained from visualization.
Whether allogeneic T cell responses are implicated in the pathogenesis of early post-HCT lung diseases. | 4 years
  This is a qualitative binary endpoint assessed by visualization.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Flerlage, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols